CLINICAL TRIAL: NCT04467489
Title: Biomarkers of Cerebral Cavernous Angioma With Symptomatic Hemorrhage (CASH)
Brief Title: Biomarkers of CASH
Status: Active, not recruiting | Type: Observational
Sponsor: University of Chicago (Other)
Collaborators: Mayo Clinic (Other); University of California, San Francisco (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Barrow Neurological Institute (Other)
Responsible Party: Sponsor
Other Study IDs: IRB20-0518; 5R01NS114552-05 (NIH)
Record Dates: First submitted 2020-07-08; First posted 2020-07-13 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Cerebral Cavernous Malformation; Cavernous Angioma; Hemorrhagic Microangiopathy
Keywords: plasma biomarker; imaging biomarker; machine learning
MeSH Terms: conditions — Hemangioma, Cavernous, Central Nervous System; Hemangioma, Cavernous | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- CA (non-CASH): Cavernous Angioma (CA) without symptomatic hemorrhage cases scheduled for evaluation by their neurology or neurosurgery teams in an inpatient or outpatient setting
  Interventions: Other: observational
- CA (CASH): Cavernous Angioma (CA) with Symptomatic Hemorrhage (SH) cases scheduled for evaluation by their neurology or neurosurgery teams in an inpatient or outpatient setting
  Interventions: Other: observational
- Young with seizure: Young (<30 years old) healthy control cohorts with seizures in the prior year
  Interventions: Other: observational
- Young without seizure: Young (<30 years old) healthy control cohorts without seizures in the prior year
  Interventions: Other: observational
- Older with HMA: Older (>50 years old) with hemorrhagic microangiopathy (HMA)
  Interventions: Other: observational
- Older without HMA: Older (>50 years old) without hemorrhagic microangiopathy (HMA)
  Interventions: Other: observational

INTERVENTIONS:
Other: observational — There is no intervention for any group in this observational study.

SUMMARY:
The project aims to develop prognostic and diagnostic blood tests for symptomatic brain hemorrhage in patients diagnosed with cavernous angiomas, a critical clinical challenge in a disease affecting more than a million Americans. We further examine whether blood biomarkers can replace or enhance the accuracy of advanced imaging in association with lesional bleeding. The project tests a novel integrational approach of biomarker development in a mechanistically defined cerebrovascular disease, with a clinically relevant context of use.

DETAILED DESCRIPTION:
Cerebral cavernous angioma (CA) is a capillary microangiopathy affecting more than a million Americans, predisposing them to a premature risk of brain hemorrhage. Fewer than 200,000 cases who have suffered a recent symptomatic hemorrhage (SH) are most likely to re-bleed again with serious clinical sequelae, and are the primary focus of therapeutic development. Genetic mechanisms of CA have been extensively studied, and consequent signaling aberrations in the neurovascular unit. These include proliferative dysangiogenesis, blood-brain barrier hyperpermeability, inflammation and immune mediated processes, anticoagulant vascular domain, and gut microbiome-driven mechanisms. Plasma levels of molecules reflecting these mechanisms and measures of vascular permeability and hemorrhage leak on magnetic resonance imaging (MRI) have been correlated with CA hemorrhage in pilot studies. It would be desirable to optimize these biomarkers to accurately diagnose CASH, to prognosticate the risk of future SH, and to monitor cases after a bleed and in response to therapy. This would influence clinical management, and select higher risk cases for clinical trials. Additional candidate biomarkers are emerging from ongoing mechanistic and differential transcriptome studies, which would be expected to further enhance the sensitivity and specificity of diagnosis and prediction of CASH. Weighed combinations of levels of plasma proteins and characteristic micro-ribonucleic acids (miRNA) may further strengthen biomarker associations. Plasma biomarkers may reflect (and potentially replace) more cumbersome and expensive imaging biomarkers for monitoring CA hemorrhage. We here assemble CA researchers and propose to deploy advanced statistical and computational biology approaches for the integration of novel candidate biomarkers. In Specific Aim 1 we assess these biomarkers in a large CA cohort to discover the best plasma biomarkers and validate them in sex, age and relevant clinical subgroups. In Specific Aim 2 we compare changes in MRI measures of vascular permeability and hemorrhage with plasma biomarkers over time. In Specific Aim 3 we query the biomarkers in non-CA subjects, to identify potential confounders in the clinical context. This project integrates analytic and computational biology expertise to develop blood tests for better CASH diagnosis and prognosis. The project tests a novel integrational approach of biomarker development in a mechanistically defined cerebrovascular disease with a relevant context of use. This approach is applicable to other neurological diseases with similar pathobiologic features.

ELIGIBILITY:
Aim 1 and 2:

Inclusion Criteria:

1. Clinical diagnosis of CA
2. age 18 or older
3. solitary or multiple
4. familial or sporadic
5. with or without prior symptoms

Exclusion Criteria:

1. Prior excision of a solitary CA lesion
2. prior stereotactic radiosurgery or any brain irradiation
3. spinal cavernoma without brain lesion
4. other brain pathology unrelated to CA (demyelinating disease, brain tumor)
5. seizures or stroke unrelated to CA in the prior year
6. current pregnancy or within 6 months postpartum
7. reluctance to undergo venipuncture or donate blood specimen, or be called for clinical follow-up for up to one year
8. homeless or incarcerated persons, or other reason a subject will be unable/unlikely to be reached for follow-up

Aim 3:

Inclusion Criteria:

1. < 30 years of age
2. one or more seizures (with or without medical therapy) in the prior year

OR

1. > 50 years of age
2. having received an MRI of the brain with SWI (susceptibility weighted imaging) sequences for any indication in the year prior to enrollment
3. No HMA on brain MRI SWI sequences

OR

1. > 50 years of age
2. having received an MRI of the brain with SWI sequences for any indication in the year prior to enrollment
3. Two or more microbleeds on SWI brain MRI sequences, adjudicated by neuroradiologist

Exclusion Criteria:

1. concurrent brain disease or structural brain pathology
2. medical illness requiring hospitalization or surgery, seizure or stroke in the prior 12 months
3. active use of prescription medications in the prior 12 months
4. current pregnancy or within 6 months postpartum
5. reluctance to undergo venipuncture or donate blood specimen

OR

1. concurrent brain disease or structural brain pathology
2. medical illness requiring hospitalization or surgery, or stroke in the prior 12 months other than seizure disorder
3. active use of prescription medications in the prior 12 months except anticonvulsants
4. current pregnancy or within 6 months postpartum
5. reluctance to undergo venipuncture or donate blood specimen

OR

1. concurrent brain disease or structural brain pathology
2. medical illness requiring hospitalization or surgery within the prior year
3. any history of stroke or epileptic seizure within the prior year
4. current pregnancy or within 6 months postpartum
5. reluctance to undergo venipuncture or donate blood specimen

OR

1. concurrent brain disease or structural brain pathology
2. medical illness requiring hospitalization or surgery within the prior year
3. any history of stroke or epileptic seizure within the prior year
4. current pregnancy or within 6 months postpartum
5. reluctance to undergo venipuncture or donate blood specimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We propose to recruit human subjects at three sites, with the project approved and coordinated by the University of Chicago Medicine (UCM) central institutional review board (IRB) and endorsed by respective IRBs at the other two enrolling sites. The study involves no more than minimal risks, discussed herein. The enrolling sites include UCM where the project will be led and where the data coordinating center (DCC) is located and all plasma biomarker assays and statistical analyses are planned, the University of California at San Francisco (UCSF), and Mayo Clinic, Rochester, MN (Mayo). UCSF and Mayo are participants in imaging biomarker validations in longitudinal follow-up of cavernous angioma with symptomatic hemorrhage (CASH) subjects in the TR Project. We project enrolling 1,040 cases during 4 years to address hypotheses in 3 Specific Aims (40 cases enrolled in Specific Aim 2 are also included among the 800 subjects addressing hypotheses of Specific Aim 1).
Sampling Method: Non-Probability Sample
Enrollment: 1040 (Estimated)
Dates: Start 2020-05-22 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Circulating Diagnostic and Prognostic Biomarkers of CASH | 5 years
  To test whether individual and combined levels of candidate plasma proteins and miRNAs can be associated with diagnosis of CASH (cross sectional) and can predict/prognosticate future SH (longitudinal) in CAs

SECONDARY OUTCOMES:
Correlation of Imaging and Plasma Biomarkers of CASH | 5 years
  To assess whether changes in QSM (quantitative susceptibility mapping) and DCEQP (dynamic contrast enhanced quantitative permeability) used as monitoring biomarkers after a SH, are reflected by changes in plasma biomarkers and miRNAs
Confounders of CASH Biomarkers | 5 years
  To assess the plasma biomarkers in non-CA young and older subjects, with and without seizures and hemorrhagic microangiopathy on MRI, to clarify potential confounders in the context of clinical use, and to motivate novel hypotheses for broader applications

CONTACTS AND LOCATIONS:
Overall Officials: Issam Awad, MD, Principal Investigator — University of Chicago
Locations (4):
- United States (4):
  - Barrow Neurological Institute at St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - University of California, San Francisco, San Francisco, California
  - The University of Chicago Medical Center, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: Yes
Within the first year, we will publish the protocol paper. At the end of the 5 year study, we will publish the data dictionary along with study findings. The expression profile data will be made publicly available no later than the date of initial publication or six months after the receipt of the final sequencing data, whichever comes first.
Supporting Information: Study Protocol, SAP
Time Frame: The expression profile data will be made publicly available no later than the date of initial publication or six months after the receipt of the final sequencing data, whichever comes first.
Access Criteria: The expression profile data will be made publicly available.

REFERENCES:
- [Derived] Girard R, Li Y, Stadnik A, Shenkar R, Hobson N, Romanos S, Srinath A, Moore T, Lightle R, Shkoukani A, Akers A, Carroll T, Christoforidis GA, Koenig JI, Lee C, Piedad K, Greenberg SM, Kim H, Flemming KD, Ji Y, Awad IA. A Roadmap for Developing Plasma Diagnostic and Prognostic Biomarkers of Cerebral Cavernous Angioma With Symptomatic Hemorrhage (CASH). Neurosurgery. 2021 Feb 16;88(3):686-697. doi: 10.1093/neuros/nyaa478. PMID 33469662